CLINICAL TRIAL: NCT00289367
Title: Randomized Prospective Study of T3 on the Incidence of Post-Operative Atrial Fibrillation in Patients Undergoing Cardiac Surgery
Brief Title: Study of T3 on the Incidence of Atrial Fibrillation in Patients Undergoing Cardiac Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Thomas and Jeanne Elmezzi Foundation (Other)
Responsible Party: Irwin Klein, North Shore University Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 05-075
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Triiodothyronine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Triiodothyronine — 0.8 mcg/kg bolus loading dose followed by a six hour infusion of 0.8 mcg/kg/6hr.
Drug: triiodothyronine — IV formulation - Triostat, 0.8 mcg/kg bolus loading dose followed by a six hour infusion of 0.8 mcg/kg/6hr.

SUMMARY:
The purpose of this project is to see whether treatment with a thyroid hormone, called triiodothyronine or T3, following open heart surgery reduces the risk of developing atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring CABG or valve repair/replacement surgery.
2. Patient must be able to provide informed consent.

Exclusion Criteria:

1. Patients less than 18 or over 85 years of age.
2. Patients less than 50kg or greater than 120kg.
3. Patients currently with endocrine disorders, excluding diabetes.
4. Patients currently with thyroid dysfunction (e.g., hyper- hyperthyroidism, goiter, Grave's disease), myxedema, or myxedema coma, even if treated.
5. Patients currently receiving thyroid replacement therapy.
6. Patients currently receiving Ketamine, levarterenol or dietary (non-food) iodine supplementation.
7. Patients who have received any investigational drugs within the previous one month or five half-lives of the drug.
8. Patients who are pregnant. Pregnancy testing will be done for women of child-bearing potential.
9. Patients currently in atrial fibrillation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2006-02; Primary Completion 2006-08 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
incidence of atrial fibrillation | during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Irwin Klein, MD, Principal Investigator — North Shore University Hospital
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States